CLINICAL TRIAL: NCT04823988
Title: Emotional, Social, Cognitive and Behavioral Sequalae of the COVID-19 Pandemic.
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000376; 000376-M
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteer
Keywords: Social Isolation; virtual; Vaccine; Anxiety; Chronic Covid; Natural History
MeSH Terms: conditions — Social Isolation; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults 18 and over: Adults 18 and over

SUMMARY:
Background:

COVID-19 has caused a high rate of deaths. The steps taken to control its spread have caused social isolation, changes in lifestyle, economic turmoil, and increased work-related stress. As a result, there has been a rise in mental and physical health problems. These burdens are particularly severe for people with a history of mental illness. Researchers want to learn more about the relationship between stressors related to COVID-19 and self-rated measures of anxiety and other variables.

Objective:

To better understand the impact of this stressful time on people s lives and families. Also, to learn the strategies people have been using to deal with the COVID-19 pandemic.

Eligibility:

Adults ages 18 and older.

Design:

This is an online study.

Participants will fill out surveys online. The surveys will ask about their mood, anxiety, medical history, substance use, and COVID-19 stressors.

Participants will complete an online task. For the task, they will stare at the center of a computer screen. When they see certain images, they will indicate the location of that image as quickly as possible.

It will take about 1.5 hours for participants to complete the surveys and tasks. They may be contacted again if additional data is needed.

Some participants may have taken part in other NIH studies. If so, their new data may be linked to their previously collected data.

DETAILED DESCRIPTION:
Study Description:

The goal of this protocol is to examine individual consequences of the COVID-19 pandemic, in the transition resolution phase with the arrival and distribution of the vaccine. Specifically, this protocol will capture the 'after-effects' of the pandemic at all levels of functioning (cognitive, emotional, social, behavioral), as well as its material impact (financial, occupational, educational). Particular attention will be directed to (1) the family structure (impact of the pandemic on adults as care-takers) (2) beliefs about and role of the introduction of the vaccine, and (3) the changes resulting from the prominent role that virtual communication has been playing in our society. Both negative and positive consequences will be probed. These effects will be carefully analyzed in function of age, gender, SES, race, family structure, psychopathology, and physical health.

This protocol is a follow-up of protocol 20MN112, titled Impact on Anxiety and Motivation of COVID-19 and Predictors of Individual Responses. Protocol 20MN112 was initiated in the early days of the pandemic (April 2020) and collects data on individual responses to the active phase of the pandemic. As we are conducting interim analyses, we have identified a number of questions to query more thoroughly, such as parenting, role of uncertainty, gender differences and the cumulative effects of environmental and personal stress. Most importantly, this ongoing protocol does not cover responses to the oncoming availability of the vaccine, and the potential 'return to normality.'

The same basic structure as protocol 20MN112 will be used: online questionnaires and cognitive task. (1) Questionnaires: We will use questionnaires to reliably gather 'explanatory' or 'predictive' measures, particularly regarding mental health and belief systems. To this aim, we will use well-normed and validated instruments (i.e., ASI, BDI, BRS, , DSM XC with substance questions, Hollingshead, Intolerance of Uncertainty scale, MASQ, Neuro QoL CFQ, PSS, PROMIS Social Isolation scale, STAI, PSWQ, LSAS, BFI). We will also adapt questionnaires to fit the specific focus on the COVID pandemic (Parent questionnaire, psychiatric history form, psychiatric history form, vaccine questionnaire, demographic questionnaire, COVID clinical mental health history, COVID adult survey, and clinical history checklist - medical). (2) Cognitive Tasks: We will continue to use a threat-biased attention task (dot-probe task), a modified version of the motivation finger-tapping task, and a standard loss aversion task. The finger-tapping task was discontinued with Amendment A. These tasks will provide objective measures of the impact of the prolonged effects of the pandemic context on cognitive function. This research will use a study website to consent, survey participants online, and the task.

Objectives:

The primary objective is to examine the impact of the long-standing threat presented by the pandemic and its associated societal changes (e.g., social isolation, financial burden) on cognitive, emotional, social, behavioral. This research will identify risk and resilience factors among study participants and provide clues for interventions tailored to individual characteristics (predictive measures).

Endpoints:

The endpoints are mental health and attention biases behavioral patterns associated with COVID-19 stressors in function of pre-existing clinical phenotype (based on retrospective measurements).

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. 18 years of age and older.
2. Able to read and write English.
3. Able to provide informed consent online using study website.

EXCLUSION CRITERIA:

1. There are no exclusion criteria for this study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample of convenience
Sampling Method: Non-Probability Sample
Enrollment: 2086 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Online self-report measures | Study date
  The primary objective is to examine the impact of COVID-19 pandemic and the precarious availability of the vaccine on mental health and cognitive function, in function of a host of factors, including parental situation, history of mental illness, demographic factors, clinical history, and other demographic variables.

SECONDARY OUTCOMES:
Comparison of questionnaire and neuroimaging data with baseline data | Study visit
  The secondary objective is to focus on participants who already completed SNFA studies prior to the pandemic, and for whom we have comprehensive screening data, and resting state MRI scans. These pre-COVID data will be used as predictors of responses to the chronic COVID-19 pandemic.

CONTACTS AND LOCATIONS:
Overall Officials: Maryland Pao, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States